CLINICAL TRIAL: NCT04208113
Title: Stress-free Everyday LiFe for Children and Adolescents REsearch (SELFCARE). A Protocol for a Cluster Randomised Trial Testing a School Teacher Training Programme to Deliver the .b Programme in Danish Schools.
Brief Title: Stress-free Everyday LiFe for Children and Adolescents REsearch
Acronym: SELFCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-051-000001/1145
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Mental Health; Children; Adolescent; Mindfulness; Stress
Keywords: School-based intervention; Population-based preventive strategy; Public health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School teacher training /.b (Experimental): The intervention is a multi-level, multi-component complex intervention. It consists of a school teacher training programme and the .b-programme to be delivered to pupils 11-15 years in the schools.
  The school teacher training programme consists of three parts: 1) the establishment of own mindfulness practice by participation in the eight week MBSR programme (2,5 hour group meeting once a week) and sustaining mindfulness with a regular formal daily practice; 2) completion of the four days .b residential course, and 3) completion of the 3x2-days seminars on relational competences and implementation issues regarding teaching .b (48 hours) The .b programme consists of well-described, weekly 40-60 minutes classroom sessions over 10 weeks. All the sessions have a specific theme, associated teachers' notes, power points and animations. The .b programme can only be delivered with fidelity by a trained .b teacher.
  Interventions: Behavioral: School teacher training /.b
- Usual practice (No Intervention): Usual practice

INTERVENTIONS:
Behavioral: School teacher training /.b — The intervention is a multi-level, multi-component complex intervention. It consists of a school teacher training programme and the .b-programme to be delivered to pupils 11-15 years in the schools.
  The school teacher training programme consists of three parts: 1) the establishment of own mindfulness practice by participation in the MBSR programme and sustaining mindfulness with a regular formal daily practice; 2) completion of the four days .b residential course, and 3) completion of the 3x2-days seminars on relational competences and implementation issues regarding teaching .b .
  The .b programme consists of well-described, weekly 40-60 minutes classroom sessions over 10 weeks. All the sessions have a specific theme, associated teachers' notes, power points and animations. The .b programme can only be delivered with fidelity by a trained .b teacher.
  Arms: School teacher training /.b

SUMMARY:
The primary aim is to evaluate the effectiveness of a profound school teacher training programme to teach a mindfulness-based programme (.b) in Danish schools on the pupils self-reported mental well-being at seven months.

The secondary aims are to evaluate i) the effectiveness of the profound school teacher training programme to teach the .b-programme in Danish schools on the pupils self-reported mental well-being post intervention (at five months).

DETAILED DESCRIPTION:
The study is a cluster randomised trial. From May 2018 - May 2019, we recruited the total of 110 Danish schools (27 schools from the Capital Region of Denmark, 18 schools from Region Zealand, 25 schools from Region of Southern Denmark, 30 schools from Central Denmark Region and 10 schools from Region of Northern Denmark).

The schools included the total of 191 school teachers for teacher training (56 teachers from the Capital Region of Denmark, 28 teachers from Region Zealand, 42 teachers from Region of Southern Denmark, 50 teachers from Central Denmark Region and 15 teachers from Region of Northern Denmark). Each included teacher will be asked to recruit a class of pupils (15-25 pupils) to test the effectiveness of the .b-programme (in total approx. 3000 pupils).

ELIGIBILITY:
Inclusion Criteria:

* All pupils in the enrolled school classes

Exclusion Criteria:

* None

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1774 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
The total difficulties score of the Strengths and Difficulties Questionnaire (SDQ)- youth self-report | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)

SECONDARY OUTCOMES:
The Strengths and Difficulties Questionnaire (SDQ)- youth self-report -subscales | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
The Strengths and Difficulties Questionnaire (SDQ)- youth self-report | 23.03.21: Seven months after baseline
  Changes in the scores among the total study population
The Strengths and Difficulties Questionnaire (SDQ)- youth self-report | 23.03.21: Five months after baseline
  Changes in the scores among the total study population
The Strengths and Difficulties Questionnaire (SDQ)- youth self-report | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) -short version | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) -short version | 23.03.21: Five months after baseline
  Change in the score among the total study population
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) -short version | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a total difficulties score>13.5
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) -short version | 23.03.21: Seven months after baseline
  Change in the score among the total study population
Brief Resilience Scale (BRS) | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Brief Resilience Scale (BRS) | 23.03.21: Five months after baseline
  Change in the score among the total study population
Brief Resilience Scale (BRS) | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Brief Resilience Scale (BRS) | 23.03.21: Seven months after baseline
  Change in the score among the total study population
School connectedness from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
School connectedness from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in the score among the total study population
School connectedness from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
School connectedness from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in the score among the total study population
Social competence from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Social competence from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in the score among the total study population
Social competence from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Social competence from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in the score among the total study population
Self-efficacy from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Self-efficacy from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in the score among the total study population
Self-efficacy from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Self-efficacy from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in the score among the total study population
Bullying items from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Bullying items from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Five months after baseline
  Change in proportions among the total study population
Bullying items from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Bullying items from the Danish student well-being questionnaire (DSWQ) | 23.03.21: Seven months after baseline
  Change in proportions among the total study population
EQ-5D-Y | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
EQ-5D-Y | 23.03.21: Five months after baseline
  Change in scores among the total study population
EQ-5D-Y | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
EQ-5D-Y | 23.03.21: Seven months after baseline
  Change in scores among the total study population
Sleep quality | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Sleep quality | 23.03.21: Five months after baseline
  Change in score among the total study population
Sleep quality | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Sleep quality | 23.03.21: Seven months after baseline
  Change in score among the total study population
Child-Adolescent Mindfulness Measure (CAMM) | 23.03.21: Five months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Child-Adolescent Mindfulness Measure (CAMM) | 23.03.21: Five months after baseline
  Change in score among the total study population
Child-Adolescent Mindfulness Measure (CAMM) | 23.03.21: Seven months after baseline
  Change in the score among the subgroup with a SDQ total difficulties score >= the 80 % percentile (23.03.21: We have chosen to identify the vulnarable group according to the standard for SDQ norms which is the >=80 % percentile. We identify per gender due to well-known differences)
Child-Adolescent Mindfulness Measure (CAMM) | 23.03.21: Seven months after baseline
  Change in score among the total study population

CONTACTS AND LOCATIONS:
Overall Officials: Lise Juul, PhD, Principal Investigator — Danish Center for Mindfulness
Locations (1):
- Danish Center for Mindfulness, Aarhus, Brabrand, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data will be shared by reasonable request, following publication of planned papers.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Juul L, Frydenberg M, Beck MS, Fjorback LO. Stress-free Everyday LiFe for Children and Adolescents REsearch (SELFCARE): a protocol for a cluster randomised trial testing a school teacher training programme to teach mindfulness (".b"). BMC Psychol. 2021 Feb 17;9(1):31. doi: 10.1186/s40359-021-00530-9. PMID 33597044